CLINICAL TRIAL: NCT05210192
Title: Sphenopalatine Ganglion Blockade With Local Analgesic in Episodic Migraine
Brief Title: Sphenopalatine Ganglion Blockade in Migraine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Gökçe Zeytin Demiral, Doctor Lecturer, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 303
Record Dates: First submitted 2021-12-03; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Episodic Migraine
MeSH Terms: interventions — Lidocaine; Solutions

STUDY DESIGN:
Intervention Model Description: Injection into the sphenopalatine ganglion of the patients in both groups will be made by entering the arcus zygomaticum and oriented at a 45 degree angle towards the opposite tooth. Injections will be made with a dental injector. The first group will be injected with 4ml of 1% lidocaine, and the second group will be injected with 4ml of 0.9% saline. Injections will be repeated weekly for the first 4 weeks, then monthly. At the end of the 1st and 3rd months of the treatment, the patients will be evaluated in the routine outpatient clinic control, and the two groups will be compared statistically by questioning the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain.
Who Masked: Participant, Investigator
Masking Description: Double-blind placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- placebo arm (Placebo Comparator): Injection into the sphenopalatine ganglion of the patients in both groups will be made by entering the arcus zygomaticum and oriented at a 45 degree angle towards the opposite tooth. Injections will be made with a dental injector. Placebo group will be injected with 4ml of 0.9% saline. Injections will be repeated weekly for the first 4 weeks, then monthly. At the end of the 1st and 3rd months of the treatment, the patients will be evaluated in the routine outpatient clinic control, and the two groups will be compared statistically by questioning the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain.
  Interventions: Drug: Placebo
- lidocaine arm (Active Comparator): Injection into the sphenopalatine ganglion of the patients in both groups will be made by entering the arcus zygomaticum and oriented at a 45 degree angle towards the opposite tooth. Injections will be made with a dental injector. Lidocaine group will be injected with 4ml of 0.1%Lidocaine. Injections will be repeated weekly for the first 4 weeks, then monthly. At the end of the 1st and 3rd months of the treatment, the patients will be evaluated in the routine outpatient clinic control, and the two groups will be compared statistically by questioning the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain.
  Interventions: Drug: Lidocaine Hydrochloride 1% Solution for Injection_#2

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 1% Solution for Injection_#2 — Injection into the sphenopalatine ganglion of the patients in both groups will be made by entering the arcus zygomaticum and oriented at a 45 degree angle towards the opposite tooth. Injections will be made with a dental injector. The first group will be injected with 4ml of 1% lidocaine. Injections will be repeated weekly for the first 4 weeks, then monthly. At the end of the 1st and 3rd months of the treatment, the patients will be evaluated in the routine outpatient clinic control, and the two groups will be compared statistically by questioning the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain.
  Arms: lidocaine arm
Drug: Placebo — Injection into the sphenopalatine ganglion of the patients in both groups will be made by entering the arcus zygomaticum and oriented at a 45 degree angle towards the opposite tooth. Injections will be made with a dental injector. The second group will be injected with 4ml of 0.9% saline. Injections will be repeated weekly for the first 4 weeks, then monthly. At the end of the 1st and 3rd months of the treatment, the patients will be evaluated in the routine outpatient clinic control, and the two groups will be compared statistically by questioning the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain.
  Arms: placebo arm

SUMMARY:
Migraine is a fairly common disease that is a leading cause of disability worldwide. 15% of the general population suffer from migraine headaches. Although there are currently many options for the treatment of acute migraine, these treatment options, such as acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDS), triptans, combinations analgesics and antiemetics, have insufficient efficacy and significant side effects. Therefore, there is a need for new treatment modalities in migraine. Sphenopalatine ganglion (SPG) block is gaining interest as an effective treatment for migraine, other headaches and facial pain syndromes.

In our study, we aimed to block the Sphenopalatine ganglion with a local anesthetic drug and compare it with the placebo control group.

DETAILED DESCRIPTION:
Between 1 May and 1 December 2021, 50 patients aged 18-50 years, who were diagnosed with episodic migraine according to ICD III criteria, who applied to the headache outpatient clinic of Afyonkarahisar Health Sciences University Medical Faculty Hospital, are planned to be included in the study. Patients with similar age, gender and disease duration will be randomly divided into 2 groups using the closed envelope method. Demographic information of the patients, chronic disease history, medications used, and duration of disease will be questioned. Before the treatment, the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain will be questioned. VAS (visual analog scale) is a scale that evaluates the severity of pain. This scale consists of numerical values between 0 and 10. 0 is considered no pain, and 10 is considered the most severe pain. Routine attack treatment of the patients will continue. Injection into the sphenopalatine ganglion of the patients in both groups will be made by entering the arcus zygomaticum and oriented at a 45 degree angle towards the opposite tooth. Injections will be made with a dental injector. The first group will be injected with 4ml of 1% lidocaine, and the second group will be injected with 4ml of 0.9% saline. Injections will be repeated weekly for the first 4 weeks, then monthly. At the end of the 1st and 3rd months of the treatment, the patients will be evaluated in the routine outpatient clinic control, and the two groups will be compared statistically by questioning the frequency of pain, the number of attacks, the severity of pain (VAS), and the duration of pain.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of episodic migraine (according to ICD-III)
* Receiving any prophylaxis treatment in the last 3 months,

Exclusion Criteria:

* Being pregnant and lactating
* Neurological and psychiatric conditions (
* Contraindications to the use of local anesthetics
* Other chronic painful conditions,
* Having a history of malignancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and Pain Level of Migraines Post-Treatment | 3-6 months after start
  The frequency and pain level of subjects' migraines will be assessed upon the conclusion of the study through surveying and comparing to previous survey data.

IPD SHARING:
Plan to Share IPD: Yes